CLINICAL TRIAL: NCT06553261
Title: Open Versus Laparoscopic Right Colectomy: Does the Initial Approach Impact on Management and Outcome in Anastomotic Leakage? A Multicenter Cohort Study
Brief Title: Anastomotic Leakage in Right Colectomy
Status: Recruiting | Type: Observational
Sponsor: Barmherzige Brüder Vienna (Other)
Collaborators: Barmherzige Brüder Salzburg (Other); Kepler University Hospital (Other); University of Salzburg (Other); Hospital Barmherzige Schwestern Vienna (Other); Medical University of Vienna (Other); University Hospital, Saarland (Other); Sigmund Freud PrivatUniversitat (Other)
Responsible Party: Principal Investigator, ILIYAN ILIEV, Dr., Barmherzige Brüder Vienna
Other Study IDs: LEAK1
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Anastomotic Leak
MeSH Terms: conditions — Anastomotic Leak | interventions — Therapeutic Irrigation; Drainage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients after laparoscopic right hemicolectomy: Patients who had undergone a laparoscopic tight colectomy and had anastomotic leak.
  Interventions: Procedure: suturing of leak, lavage, drainage; Procedure: Formation of a new anasthomosis; Procedure: Fecal diversion
- Patients after open right hemicolectomy: Patients who had undergone a laparoscopic tight colectomy and had anastomotic leak.
  Interventions: Procedure: suturing of leak, lavage, drainage; Procedure: Formation of a new anasthomosis; Procedure: Fecal diversion

INTERVENTIONS:
Procedure: suturing of leak, lavage, drainage — Operative suturing of the leak, lavage, drainage within a revision surgery.
Procedure: Formation of a new anasthomosis — Operative resection of the old leaking anastomosis and formation of a new one.
Procedure: Fecal diversion — Formation of a deviating stoma.

SUMMARY:
Data of patients undergoing elective right colectomy for benign and malignant disease using an open or laparoscopic approach are to be collected in seven colorectal units among Austria for the period between January 2010 and December 2019. Demographic, peri- and postoperative data of patients were analyzed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign or malignant diseases in the right portion of the colon.
* elective surgery

Exclusion Criteria:

* emergent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with benign or malignant diseases in the right colon.
Sampling Method: Probability Sample
Enrollment: 3446 (Estimated)
Dates: Start 2024-08-12 (Estimated); Primary Completion 2024-10-12 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome | 2010-2019
  Survival or death

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Dauser, Assoc. Prof., Principal Investigator — Krankenhaus der Barmherzigen Brüder Vienna
Locations (1):
- Krankenhaus der Barmherzigen Brüder, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided